CLINICAL TRIAL: NCT02317939
Title: Home Monitoring of Patients With Rheumatoid Arthritis - an eHealth Development Study
Acronym: ELECTOR_I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Gudbergsen (Other)
Collaborators: Charles University, Czech Republic (Other); Region Capital Denmark (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, EU project coordinator, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100.01
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- online instruction at followup visits (Experimental): patients in this group will be subjected to view video instructions online prior to performing the follow-up joint scoring at home
  Interventions: Other: instruction
- standard baseline instruction (Active Comparator): after the initial training patients in this group will not be subjected to any subsequent instructions prior to performing the follow-up joint scoring at home
  Interventions: Other: standard baseline instruction

INTERVENTIONS:
Other: instruction — online instruction tutorials at followup visits
  Arms: online instruction at followup visits
Other: standard baseline instruction — self-guidance at followup visits
  Arms: standard baseline instruction

SUMMARY:
A two-step multi-centre study with 240 rheumatoid arthritis patients.

DETAILED DESCRIPTION:
A two-step multi-centre study containing:

A test-retest study including 180 patients filling in questionnaires and performing joint assessments to assess reliability of patient generated data

AND

An agreement study focusing on questionnaires and joint assessments performed by 60 patients, a medical student, a physician and by an ultrasound-examinator assessing agreement between the four assessors

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA ≥ 12 months
* DAS28-CRP < 5,1

Exclusion Criteria:

* Dementia or other linguistic/cognitive/physical deficiency that prevents participation
* Vision impairment that prevents the use of the devices and computer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Intrarater reliability of DAS28 done by patients | Baseline

SECONDARY OUTCOMES:
Interrater agreement of DAS28CRP | Baseline
Intrarater reliability of joints counts performed by patients | Baseline
Intrarater reliability of joint scores performed by patients | 8 weeks
Inter- and intrarater realiabilty of DAS38 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hennning Bliddal, MD, DMSc, Study Director — Parker RI; Henrik R Gudbergsen, MD, PhD, Principal Investigator — Parker RI
Locations (1):
- Department of Rheumatology, Frederiksberg, Capital Region, Denmark

REFERENCES:
- [Derived] Skougaard M, Bliddal H, Christensen R, Ellegaard K, Nielsen SM, Zavada J, Oreska S, Krogh NS, Holm CC, Hetland ML, Vencovsky J, Rogind H, Taylor PC, Gudbergsen H. Patients with Rheumatoid Arthritis Acquire Sustainable Skills for Home Monitoring: A Prospective Dual-country Cohort Study (ELECTOR Clinical Trial I). J Rheumatol. 2020 May 1;47(5):658-667. doi: 10.3899/jrheum.181362. Epub 2019 Aug 15. PMID 31416921